CLINICAL TRIAL: NCT01143870
Title: Examining Ways to Increase Patient Understanding of Diabetes Control and Disease Severity Through Reinterpretation of Hemoglobin A1C Values With the Goal of Improved Diabetes Control
Brief Title: New Ways to Help Patients Improve Their Diabetes Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 811355
Record Dates: First submitted 2010-05-17; First posted 2010-06-14 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hemoglobin A1C (Other): Diabetes control related to patients using standard hemoglobin A1C
  Interventions: Other: "Diabetes Report Card"
- Face (Experimental): Face expressing emotion used to depict diabetes control
  Interventions: Other: "Diabetes Report Card"
- Letter grade (Experimental): Letter grade used to express diabetes control
  Interventions: Other: "Diabetes Report Card"

INTERVENTIONS:
Other: "Diabetes Report Card" — Enrolled participants will receive an individualized "diabetes report card" which depicts their current level of diabetes control in one of three ways--hemoglobin A1C, face, or letter grade.

SUMMARY:
The percent of glycosylated hemoglobin, also known as a hemoglobin A1C value, is the standard way that clinicians assess a patient's diabetes control. Numerous studies have shown that maintaining a hemoglobin A1C value less than 7% is associated with lower rates of diabetes-related complications. Clinicians use this value to determine whether a patient with diabetes requires changes in their disease management. The main problem with this practice is that many patients do not understand what this number means. The goal of this project is to examine ways to make feedback about glycemic control easier for patients to understand. The hope is that improved patient understanding will result in an improvement in diabetic control and thus a reduction in disease-associated complications. Patients with a diagnosis of diabetes and a hemoglobin A1C value greater than 8% within the preceding three months will be eligible for the study. Pregnant women will be excluded. Given the nature of the intervention we will also exclude patients with cognitive deficits. In this study, patients will be randomized to three groups. The first group with be told their HgbA1C value only, the second group will be told a letter grade interpretation of that value, and the third group will be shown a face. The face emotions will range from happy to sad reflecting the level of control. The main outcome will be trend in hemoglobin A1C values over time. Secondary outcomes will include patient understanding of disease state and the number of hemoglobin A1C values checked following the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 18 with diabetes mellitus listed as a problem list or in their past medical history on their electronic medical record who have a hemoglobin A1C value greater than 8% within three months of study enrollment.

Exclusion Criteria:

1. Pregnant patients
2. Illiterate patients
3. Patients with known cognitive deficits affecting ability to participate in study
4. Any current participants in another active research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Volpp, M.D., PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Gopalan A, Tahirovic E, Moss H, Troxel AB, Zhu J, Loewenstein G, Volpp KG. Translating the hemoglobin A1C with more easily understood feedback: a randomized controlled trial. J Gen Intern Med. 2014 Jul;29(7):996-1003. doi: 10.1007/s11606-014-2810-4. Epub 2014 Feb 25. PMID 24567202

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Received information on diabetes control using the standard hemoglobin A1c value
- Letter Grades: Received information on diabetes control translated into a letter grade, ranging from A-F
- Faces: Received information on diabetes control translated into a emoticon, ranging from smiling to crying
Period: Overall Study
Arm/Group | Control | Letter Grades | Faces
Started | 58 | 58 | 61
Post-intervention Survey | 53 | 50 | 61
Had Available 6-month A1C | 27 | 29 | 31
A1C Imputed | 31 | 29 | 30
Completed | 58 | 58 | 61
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Letter Grades | Faces | Total
Number analyzed (Participants) | 58 | 58 | 61 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (3.3) | 57.8 (3.1) | 55 (3.5) | 56.4 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 45 | 44 | 130
  Male | 17 | 13 | 17 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 48 | 50 | 48 | 146
  White | 2 | 2 | 4 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 8 | 6 | 9 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent of Glycosylated Hemoglobin 6 Months Following Enrollment
Time Frame: 6 months from enrollment
Measure: Mean (Standard Error); unit: Percent of glycosylated hemoglobin
Arm/Group | Control | Letter Grades | Faces
Number analyzed (Participants) | 58 | 58 | 61
Percent of glycosylated hemoglobin | -0.74 (0.37) | -0.55 (0.3) | -0.89 (0.3)

2. Secondary Outcome: Change in Patient Understanding of Disease State
Description: Change in patient understanding of disease state as assessed by questionnaire administered pre- and post-intervention.
Time Frame: 2 weeks on average
Reporting Status: Not Posted

3. Secondary Outcome: The Number of Hemoglobin A1C Values Checked During 6 Month Study Period
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Change in Hemoglobin A1C Over 12 Months From Enrollment
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Control | Letter Grades | Faces
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/58 | 0/61
Other Adverse Events (participants affected / at risk) | 0/58 | 0/58 | 0/61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No